CLINICAL TRIAL: NCT04229823
Title: Natural History of Oculomotor Neurophysiology in Ataxic and Pre-ataxic Carriers of Machado-Joseph Disease/Spinocerebellar Ataxia Type 3 (SCA3/MJD)
Brief Title: Natural History of Oculomotor Neurophysiology in Ataxic and Pre-ataxic Carriers of SCA3/MJD
Acronym: BIGPRO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-0015
Record Dates: First submitted 2020-01-07; First posted 2020-01-18 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Spinocerebellar Ataxia Type 3; Machado-Joseph Disease
Keywords: Machado-Joseph Disease; Spinocerebellar Ataxia Type 3; SCA3; Biomarker; Natural history; Video-oculography; Eye movement; Surrogate biomarker; Oculomotor neurophysiology
MeSH Terms: conditions — Machado-Joseph Disease | interventions — Genotype

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ataxic carriers: Subjects with a CAG repeat expansion on ATXN3 and Scale for Assessment and Rating of Ataxia (SARA) of 3 points or more.
  Interventions: Diagnostic Test: Video-oculography; Diagnostic Test: Clinical Scales
- Pre-ataxic carriers: Subjects with a CAG repeat expansion on ATXN3 and Scale for Assessment and Rating of Ataxia (SARA) of less than 3 points.
  Interventions: Diagnostic Test: Video-oculography; Diagnostic Test: Clinical Scales; Diagnostic Test: Genotyping
- Related controls: Subjects without a CAG repeat expansion on ATXN3, but with a first degree relative affected by the disease.
  Interventions: Diagnostic Test: Video-oculography; Diagnostic Test: Clinical Scales; Diagnostic Test: Genotyping

INTERVENTIONS:
Diagnostic Test: Video-oculography — Eye movement parameters will be measured in all of the subjects using video-oculography device (EyeSeeCam, InterAcoustics). Measurement sessions consist of the study subject wearing a goggle attached to a camera that detects the pupil and eye position and velocity. Evaluation start with vestibulo-ocular reflex testing, with video head impulse test. Afterwards, saccades, smooth pursuit and fixation are evaluated.
Diagnostic Test: Clinical Scales — All subjects are examined by an investigator in order to score clinical scales for ataxia, including Scale for the Assessment and Rating of Ataxia (SARA), International Co-operative Rating Scale (ICARS), Neurological Examination Scale for SCA (NESSCA), Inventory of Non-ataxia Symptoms (INAS), SCA Functional Index (SCAFI) and Composite Cerebellar Functional Severity Score (CCFS).
Diagnostic Test: Genotyping — Individuals at 50% risk (offspring of subjects with molecular diagnosis of SCA3/MJD) will be genotyped in a double-blind manner so that they can be divided into pre-ataxic carriers and related controls (non carriers)
  Groups: Pre-ataxic carriers; Related controls

SUMMARY:
The study will consist of a prospective observation of subjects in a natural history design. Disease progression will be monitored through clinical scales and video-oculography. Participants will be stratified in three groups: ataxic carriers, pre-ataxic carriers and non-carriers (controls). The following clinical scales will be applied in all subjects at baseline and at months 12 and 24: SARA, SCAFI, CCFS, NESSCA, INAS and ICARS. Oculomotor function will be registered using video-oculography (EyeSeeCam, InterAcoustics) at the same time points. Progression rates, effect sizes and responsiveness to change will be established for all parameters and results will be compared between candidate biomarkers.

DETAILED DESCRIPTION:
Spinocerebellar ataxia type 3, also called Machado-Joseph disease (SCA3/MJD), is an autosomal dominant neurodegenerative disorder caused by a CAG expansion (CAGexp) on ATXN3. Over 20 years after the identification of the causal mutation, no form of prevention or treatment for this incapacitating condition was discovered. Similarly to other polyglutamine (polyQ) diseases, SCA3/MJD has a slow progression. Changes detected by clinical scales are small and, therefore, long intervals are needed to document disease progression. Clinical trials using clinical scales as primary outcomes should be very long, what makes them hardly feasible. In this context, the discovery of disease biomarkers is of utmost importance. Biomarkers associated with disease progression and/or with therapeutic intervention might be more easily verified than the changes measured by clinical scales. Seminal studies have demonstrated that oculomotor alterations and vestibulo-ocular reflex (VOR) impairment may be present even during presymptomatic periods. Our primary hypothesis is eye movement parameters including VOR, saccades, smooth pursuit and fixation measured by video-oculography could be biomarkers of SCA3/MJD disease progression. Besides that, the investigators aim to test if the candidate biomarkers present changes before disease-onset and if their responsiveness will be better than those of clinical scales, with more noticeable variations during a shorter period of time. The study will consist of a prospective observation of subjects in a natural history design. The investigators will monitor disease progression of the CAGexp carriers through clinical scales and video-oculography. At least 75 adult subjects from Rio Grande do Sul will be invited to participate in the study, and at least 50 of the participants will be asymptomatic subjects, at 50% risk of carrying the mutation. The study design will allow the subjects who wanted and the evaluators to stay blinded to subjects' genotypes. Participants will be stratified in three groups: ataxic carriers, pre-ataxic carriers and non-carriers (controls). Genotypes will be recorded separately to guarantee double blindness. For every pre-ataxic carrier, time until the disease-onset will be estimated by an equation previously built, in which individual age and CAGexp are the determinants. The following clinical scales will be applied in all subjects at baseline and at months 12 and 24: SARA, SCAFI, CCFS, NESSCA, INAS and ICARS. Oculomotor function will be registered in video and analyzed using the EyeSeeCam device. Progression rates of all variables will be estimated by mixed models, including as covariates age, groups and their interactions. Progression rates, effect sizes and responsiveness to change will be established for all parameters and results will be compared between candidate biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with molecular diagnosis of SCA3/MJD
* Individuals at 50% risk of inheriting SCA3/MJD mutation without any clinical manifestation

Exclusion Criteria:

* Other diagnosed neurological or vestibular condition
* Dyschromatopsia
* Refusal to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with molecular diagnosis of SCA3/MJD will be recruited from the Medical Genetics Service database of Hospital de Clínicas de Porto Alegre, Brazil, by telephone calls or by invitation in the outpatient clinic. First degree relatives of these subjects at 50% risk of carrying the mutation will also be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Change in vestibulo-ocular reflex gain regression slope (VORr) | 24 months
  Gain (Eye velocity/Head velocity)
Change in vertical smooth pursuit gain | 24 months
  Regression slope of eye velocity versus target velocity during vertical smooth pursuit task
Change in slow-phase velocity of gaze evoked nystagmus (SPV-GE) | 24 months
  Degrees/second
Change in the slope of peak duration versus amplitude of volitional vertical saccades | 24 months
  egression slope between peak duration and saccade amplitude during volitional vertical saccades
Change in the slope of peak duration versus amplitude of reflexive vertical saccades | 24 months
  Regression slope between peak duration and saccade amplitude during reflexive vertical saccades
Change in slow-phase velocity of central nystagmus (SPV-C) | 24 months
  Degrees/second
Change in Neurological Examination Score for Spinocerebellar Ataxia (NESSCA) | 24 months
  Neurological examination score, varying between 0 and 40. Score increases with disease severity.
Change in SCA Functional Index (SCAFI) | 24 months
  Composite score. Score decreases with disease severity.
Change in International Cooperative Ataxia Rating Scale (ICARS) | 24 months
  Absolute score, varying between 0 and 100. Score increases with disease severity.
Change in Inventory of Non-Ataxia Symptoms (INAS) count | 24 months
  Scale varying between 0 and 16. Score increases with disease severity.
Change in Composite Cerebellar Functional Severity Score (CCFS) | 24 months
  Composite score. Score increases with disease severity.

SECONDARY OUTCOMES:
Change in horizontal smooth pursuit gain | 24 months
  Gain (Eye velocity/Target velocity)
Change in reflexive vertical saccade velocity (RVSV) | 24 months
  Degrees/second
Change in volitional vertical saccade velocity (VVSV) | 24 months
  Degrees/second

CONTACTS AND LOCATIONS:
Overall Officials: Laura Jardim, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Universidade Federal do Rio Grande do Sul, Porto Alegre, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will be done via direct contact with the Principal Investigator in order to preserve individual participants identities
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will become available after final statistical analysis and data publishing via direct contact with principal investigator
Access Criteria: Investigators and researchers of the area

REFERENCES:
- See also: BIGPRO study website — https://bigpro.webnode.com/